CLINICAL TRIAL: NCT02713087
Title: Influence of Vasopressors on Brain Oxygenation and Microcirculation in Anesthetized Patients With Cerebral Tumors
Brief Title: Vasopressor Effects in Anesthetized Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vasobrain01
Record Dates: First submitted 2016-02-10; First posted 2016-03-18 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2016-10

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Ephedrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ephedrine (Active Comparator)
  Interventions: Drug: Ephedrine
- Phenylephrine (Active Comparator)
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Ephedrine — Infusion of Ephedrine 2mg/ml until MAP above 60 mmHg or until MAP has raised 20%
  Arms: Ephedrine
Drug: Phenylephrine — Infusion of Phenylephrine 0,1mg/ml until MAP above 60 mmHg or until MAP has raised 20%
  Arms: Phenylephrine

SUMMARY:
Project title: Influence of Vasopressors on Brain Oxygenation and Microcirculation in Anesthetized Patients with Cerebral Tumors

Sponsor-investigator: Klaus Ulrik Koch M.D.

Sponsor: Department of Anesthesia Aarhus University Hospital, Nørrebrogade 44, 8000 Aarhus C, Denmark

Objective:

To investigate whether phenylephrine and ephedrine causes different alterations in microcirculation and oxygenation, as measured with MRI and PET, in anesthetized patients with brain tumors. Using MRI and PET, the study will assess whether there is a difference in deoxyhemoglobin concentration (Bold signal), CTTH, cerebral blood flow (CBF) and cerebral metabolic rate of oxygen (CMRO2) between ephedrine and phenylephrine

Method:

Double blinded controlled randomized clinical trial. Either phenylephrine or ephedrine are infused intravenously under general anesthesia. MRI is performed in 20 patients before and after infusion. PET/CT is performed in 20 patients before and after infusion. BIS and NIRS monitoring will be used in either scanner. After scanning patients are transported to the operating theatre and the craniotomy is performed. After removal of the bone flap subdural ICP is measured and recorded.

MRI to analyze CBF, CTH, max.CMRO2, maxOEF, CBV and grey-scale ADC before and after ephedrine and phenylephrine. PET/CT to analyze CBF and CMRO2 before and after ephedrine and phenylephrine and calculation of OEF. During each PET/CT scan session oxygen saturation and hemoglobin concentration is measured.

Data from the proposed studies will add substantial new knowledge to the investigators current understanding of the effects of vasopressors on cerebral circulation. This information will aid the neuroanesthesiologist, neurointensivist and the neurosurgeon in the choice of the optimal method to manage cerebral perfusion pressure during craniotomy for brain tumor.

DETAILED DESCRIPTION:
Background:

During brain tumor surgery the main objective for the neuroanesthesiologist is to maintain a low intracranial pressure (ICP) and a sufficient cerebral perfusion pressure (CPP) (CPP = mean arterial blood pressure [MABP] - ICP) to ensure adequate cerebral oxygenation. Brain tumors are often associated with edema and increased ICP and a specific recommendation for CPP thresholds during brain tumor surgery does not exist. In daily practice vasopressors are used to increase MABP to maintain a CPP between 50-70 mmHg in accordance with current guidelines for management of patients with traumatic brain pathology.

However, recent studies show that arterial blood pressure correlates only poorly with microcirculatory flow. Elevation of blood pressure may result in reduced capillary perfusion and oxygen delivery despite reaching resuscitation end-points with CPP within 50-70 mmHg. This is supported by an experimental study demonstrating vasopressor-induced mismatch between cerebral perfusion and oxygenation, possibly due to microvascular heterogeneity, as suggested by the authors. In addition, recent studies in healthy anesthetized subjects demonstrate that, despite an increase in MABP, cerebral oxygenation simultaneously decreases after phenylephrine but remains unchanged after administration of ephedrine. Thus, increasing CPP with vasopressors may lead to paradoxical microcirculatory response with vasopressor-induced tissue hypo-perfusion and hindered tissue oxygenation.

Brain microcirculation is the primary site of oxygen exchange. The investigators have recently proposed that red blood cell capillary transit time heterogeneity (CTTH) may affect tissue oxygen tension in patients with ischemic stroke, subarachnoid hemorrhage and traumatic brain injury. According to this theory capillary compression due to edema and elevated ICP may cause redistribution of capillary flows into patterns with functional shunting of oxygenated blood through the cerebral capillary bed. This capillary dysfunction may further hinder oxygen diffusion into cerebral tissue and ultimately cause cerebral ischemic damage. The dissimilar effects of phenylephrine and ephedrine on cerebral oxygenation may be caused by a different influence on brain capillary perfusion or alternated CTTH. Currently there are no studies available on the effects of commonly used vasopressors on brain microcirculation and oxygenation in patients undergoing craniotomy for brain tumors.

Hypothesis:

The use of phenylephrine is associated with a reduction in brain oxygenation and microcirculation compared to ephedrine in anesthetized patients with brain tumors.

Specifically the investigators hypothesize that:

1. In peritumoral areas phenylephrine is associated with a local increase in CBF, increased CTTH, decreased oxygen extraction fraction and increase in the BOLD signal compared to ephedrine
2. Phenylephrine is associated with a reduction in oxygen extraction fraction (OEF) compared to ephedrine

Materials and methods:

Overall Study design:

Double blinded controlled randomized clinical trial.

Studies:

Study 1 (MRI study). 20 patients are randomized to infusion of either ephedrine or phenylephrine until MAP >60 mmHg

Study 2 (PET study). 20 patients are randomized to infusion of either ephedrine or phenylephrine until MAP >60mmHg

MRI and PET measurements are performed after induction of general anesthesia with propofol and remifentanil. The MRI or PET sequence is then performed before administration of study-drug and again after the infusion of either phenylephrine or ephedrine results in MAP > 60mmHg. Depth of anesthesia is monitored with BIS in both studies to ensure equal level of anesthetic depth in the two groups. NIRS is monitored in both studies to compare measurements of brain oxygenation determined by PET/CT. NIRS measurements are not possible during MR scan and will be measured either before or after the scan. BIS and NIRS are registered in each patients case report form (CRF). After the MRI/PET study the patient is transported to the operating theatre and the craniotomy is performed. After removal of the bone-flap, subdural ICP is measured and recorded as previously described.

The overall experimental setup is the same for the two studies. The patient is anesthetized and MRI or PET is performed before and after administration of a study-drug. The specific MRI and PET protocols are mentioned below

* MRI protocol
* Conventional MRI sequences on a high quality research scanner
* Diffusion-weighted MRI incl. diffusion kurtosis imaging
* Perfusion-weighted MRI before and after ephedrine or phenylephrine, respectively
* The duration of the entire MRI scan is estimated to 60 min. Two and a half standard doses of gadolinium MRI contrast are administered ( 0.25 mmol/kg).
* PET protocol
* Cerebral Blood Flow (CBF): 500 MBq of [15O]H2O is injected intravenously. At injection a three minute PET image acquisition of the brain is started together with arterial blood sampling (also three minutes) with an automated blood radioactivity sampler that draws 7 ml blood per minute. The PET acquisition is done on a Siemens High Resolution Research Tomograph (HRRT) in list mode.
* Cerebral Metabolic Rate of Oxygen (CMRO2): 1000 MBq of [15O]O2 is inhaled and immediately exhaled. At inhalation PET acquisition and blood sampling are performed with protocols identical to CBF.
* During each scan session oxygen saturation and haemoglobin concentration will be measured.

Physiological parameters (blood pressure and ICP) are documented in the CRF corresponding to each patient. BIS and NIRS data are stored on a portable computer and subjected to offline analysis. Parametric and non-parametric statistics will be used to compare MRI and PET. Physiological data will be recorded during stimulation with study-drugs. The sample size is based on previous publications where a MRI protocol was performed before and after drug administration in anesthetized patients. The exact form of applied statistics are not yet decided. This kind of study with new parameters from MRI and PET has never been done and statistical help will be consulted along the process.

Perspectives:

Data from the proposed studies will add to the investigators understanding of the cerebral microcirculation and its importance for brain oxygenation in patients of different age and comorbidity. Meanwhile, the study will provide new insights into the effects of vasopressors on the cerebral circulation. The study will thus provide direct observations for the investigators recent efforts to understand the role of the microcirculation in neurological disorders, and help the investigators chose the optimal method to manage CPP during craniotomy for brain tumor.

These insights may have implications for the future management of increased intracranial pressure and CPP after TBI and SAH.

Applicant´s part in the research:

Applicant Klaus Ulrik Koch is sponsor-investigator on this study and the responsible person of finishing the PhD thesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for supine-positioned elective craniotomy for supratentorial malignant and non-malignant brain tumors 3 cm or larger (measured as the largest diameter in any plane on MR images)
* ASA (American Society of Anesthesiologist) status 1-3 (27)
* Written informed consent from participating patients

Exclusion Criteria:

* Age younger than 18 yrs. or older than 75 yrs.
* Pregnancy or nursing (negative pregnancy blood test)
* History of allergic reactions to phenylephrine or ephedrine
* eGFR < 60ml/min/1.73m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Capillary Transit Time Heterogeneity | 4 Years

SECONDARY OUTCOMES:
Cerebral Metabolic Rate of Oxygen | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Leif Oestergaard, Professor, Study Director — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen M, Bundgaard H, Cold GE. Craniotomy for supratentorial brain tumors: risk factors for brain swelling after opening the dura mater. J Neurosurg. 2004 Oct;101(4):621-6. doi: 10.3171/jns.2004.101.4.0621. PMID 15481716
- [Background] Rasmussen M, Juul N, Christensen SM, Jonsdottir KY, Gyldensted C, Vestergaard-Poulsen P, Cold GE, Ostergaard L. Cerebral blood flow, blood volume, and mean transit time responses to propofol and indomethacin in peritumor and contralateral brain regions: perioperative perfusion-weighted magnetic resonance imaging in patients with brain tumors. Anesthesiology. 2010 Jan;112(1):50-6. doi: 10.1097/ALN.0b013e3181c38bd3. PMID 19952725
- [Background] Rasmussen M, Ostergaard L, Juul N, Gyldensted C, Poulsen PV, Cold GE. Do indomethacin and propofol cause cerebral ischemic damage? Diffusion-weighted magnetic resonance imaging in patients undergoing craniotomy for brain tumors. Anesthesiology. 2004 Oct;101(4):872-8. doi: 10.1097/00000542-200410000-00011. PMID 15448519
- [Background] Dubin A, Pozo MO, Casabella CA, Palizas F Jr, Murias G, Moseinco MC, Kanoore Edul VS, Palizas F, Estenssoro E, Ince C. Increasing arterial blood pressure with norepinephrine does not improve microcirculatory blood flow: a prospective study. Crit Care. 2009;13(3):R92. doi: 10.1186/cc7922. Epub 2009 Jun 17. PMID 19534818
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. XIV. Hyperventilation. J Neurotrauma. 2007;24 Suppl 1:S87-90. doi: 10.1089/neu.2007.9982. No abstract available. PMID 17511553
- [Background] Boerma EC, Ince C. The role of vasoactive agents in the resuscitation of microvascular perfusion and tissue oxygenation in critically ill patients. Intensive Care Med. 2010 Dec;36(12):2004-18. doi: 10.1007/s00134-010-1970-x. Epub 2010 Sep 2. PMID 20811874
- [Background] Sahuquillo J, Amoros S, Santos A, Poca MA, Panzardo H, Dominguez L, Pedraza S. Does an increase in cerebral perfusion pressure always mean a better oxygenated brain? A study in head-injured patients. Acta Neurochir Suppl. 2000;76:457-62. doi: 10.1007/978-3-7091-6346-7_95. PMID 11450067
- [Background] Hahn GH, Hyttel-Sorensen S, Petersen SM, Pryds O, Greisen G. Cerebral effects of commonly used vasopressor-inotropes: a study in newborn piglets. PLoS One. 2013 May 20;8(5):e63069. doi: 10.1371/journal.pone.0063069. Print 2013. PMID 23700412
- [Background] Nissen P, Brassard P, Jorgensen TB, Secher NH. Phenylephrine but not ephedrine reduces frontal lobe oxygenation following anesthesia-induced hypotension. Neurocrit Care. 2010 Feb;12(1):17-23. doi: 10.1007/s12028-009-9313-x. PMID 19957053
- [Background] Meng L, Cannesson M, Alexander BS, Yu Z, Kain ZN, Cerussi AE, Tromberg BJ, Mantulin WW. Effect of phenylephrine and ephedrine bolus treatment on cerebral oxygenation in anaesthetized patients. Br J Anaesth. 2011 Aug;107(2):209-17. doi: 10.1093/bja/aer150. Epub 2011 Jun 3. PMID 21642644
- [Background] Soeding PF, Hoy S, Hoy G, Evans M, Royse CF. Effect of phenylephrine on the haemodynamic state and cerebral oxygen saturation during anaesthesia in the upright position. Br J Anaesth. 2013 Aug;111(2):229-34. doi: 10.1093/bja/aet024. Epub 2013 Mar 21. PMID 23518801
- [Background] Jespersen SN, Ostergaard L. The roles of cerebral blood flow, capillary transit time heterogeneity, and oxygen tension in brain oxygenation and metabolism. J Cereb Blood Flow Metab. 2012 Feb;32(2):264-77. doi: 10.1038/jcbfm.2011.153. Epub 2011 Nov 2. PMID 22044867
- [Background] Ostergaard L, Jespersen SN, Mouridsen K, Mikkelsen IK, Jonsdottir KY, Tietze A, Blicher JU, Aamand R, Hjort N, Iversen NK, Cai C, Hougaard KD, Simonsen CZ, Von Weitzel-Mudersbach P, Modrau B, Nagenthiraja K, Riisgaard Ribe L, Hansen MB, Bekke SL, Dahlman MG, Puig J, Pedraza S, Serena J, Cho TH, Siemonsen S, Thomalla G, Fiehler J, Nighoghossian N, Andersen G. The role of the cerebral capillaries in acute ischemic stroke: the extended penumbra model. J Cereb Blood Flow Metab. 2013 May;33(5):635-48. doi: 10.1038/jcbfm.2013.18. Epub 2013 Feb 27. PMID 23443173
- [Background] Ostergaard L, Aamand R, Karabegovic S, Tietze A, Blicher JU, Mikkelsen IK, Iversen NK, Secher N, Engedal TS, Anzabi M, Jimenez EG, Cai C, Koch KU, Naess-Schmidt ET, Obel A, Juul N, Rasmussen M, Sorensen JC. The role of the microcirculation in delayed cerebral ischemia and chronic degenerative changes after subarachnoid hemorrhage. J Cereb Blood Flow Metab. 2013 Dec;33(12):1825-37. doi: 10.1038/jcbfm.2013.173. Epub 2013 Sep 25. PMID 24064495
- [Background] Ostergaard L, Engedal TS, Aamand R, Mikkelsen R, Iversen NK, Anzabi M, Naess-Schmidt ET, Drasbek KR, Bay V, Blicher JU, Tietze A, Mikkelsen IK, Hansen B, Jespersen SN, Juul N, Sorensen JC, Rasmussen M. Capillary transit time heterogeneity and flow-metabolism coupling after traumatic brain injury. J Cereb Blood Flow Metab. 2014 Oct;34(10):1585-98. doi: 10.1038/jcbfm.2014.131. Epub 2014 Jul 23. PMID 25052556
- [Background] Petersen KD, Landsfeldt U, Cold GE, Petersen CB, Mau S, Hauerberg J, Holst P, Olsen KS. Intracranial pressure and cerebral hemodynamic in patients with cerebral tumors: a randomized prospective study of patients subjected to craniotomy in propofol-fentanyl, isoflurane-fentanyl, or sevoflurane-fentanyl anesthesia. Anesthesiology. 2003 Feb;98(2):329-36. doi: 10.1097/00000542-200302000-00010. PMID 12552189
- [Background] Cold GE, Tange M, Jensen TM, Ottesen S. "Subdural' pressure measurement during craniotomy. Correlation with tactile estimation of dural tension and brain herniation after opening of dura. Br J Neurosurg. 1996 Feb;10(1):69-75. doi: 10.1080/02688699650040548. PMID 8672261
- [Background] Ostergaard L, Weisskoff RM, Chesler DA, Gyldensted C, Rosen BR. High resolution measurement of cerebral blood flow using intravascular tracer bolus passages. Part I: Mathematical approach and statistical analysis. Magn Reson Med. 1996 Nov;36(5):715-25. doi: 10.1002/mrm.1910360510. PMID 8916022
- [Background] Mouridsen K, Hansen MB, Ostergaard L, Jespersen SN. Reliable estimation of capillary transit time distributions using DSC-MRI. J Cereb Blood Flow Metab. 2014 Sep;34(9):1511-21. doi: 10.1038/jcbfm.2014.111. Epub 2014 Jun 18. PMID 24938401
- [Background] Hansen B, Lund TE, Sangill R, Jespersen SN. Experimentally and computationally fast method for estimation of a mean kurtosis. Magn Reson Med. 2013 Jun;69(6):1754-60. doi: 10.1002/mrm.24743. Epub 2013 Apr 15. PMID 23589312
- [Background] Blomqvist G. On the construction of functional maps in positron emission tomography. J Cereb Blood Flow Metab. 1984 Dec;4(4):629-32. doi: 10.1038/jcbfm.1984.89. PMID 6334095
- [Background] Ohta S, Meyer E, Fujita H, Reutens DC, Evans A, Gjedde A. Cerebral [15O]water clearance in humans determined by PET: I. Theory and normal values. J Cereb Blood Flow Metab. 1996 Sep;16(5):765-80. doi: 10.1097/00004647-199609000-00002. PMID 8784222
- [Background] Ohta S, Meyer E, Thompson CJ, Gjedde A. Oxygen consumption of the living human brain measured after a single inhalation of positron emitting oxygen. J Cereb Blood Flow Metab. 1992 Mar;12(2):179-92. doi: 10.1038/jcbfm.1992.28. PMID 1548291
- [Background] Radiation dose to patients from radiopharmaceuticals (addendum 2 to ICRP publication 53). Ann ICRP. 1998;28(3):1-126. doi: 10.1016/s0146-6453(99)00006-8. PMID 10840563
- [Background] Mak PH, Campbell RC, Irwin MG; American Society of Anesthesiologists. The ASA Physical Status Classification: inter-observer consistency. American Society of Anesthesiologists. Anaesth Intensive Care. 2002 Oct;30(5):633-40. doi: 10.1177/0310057X0203000516. PMID 12413266
- [Background] Ngwenya LB, Chiocca EA. Editorial: postoperative ischemia. J Neurosurg. 2013 Apr;118(4):799-800; discussion 800. doi: 10.3171/2012.8.JNS121410. Epub 2013 Feb 1. No abstract available. PMID 23373805
- [Derived] Koch KU, Tietze A, Aanerud J, Oettingen GV, Juul N, Sorensen JCH, Nikolajsen L, Ostergaard L, Rasmussen M. Effect of ephedrine and phenylephrine on brain oxygenation and microcirculation in anaesthetised patients with cerebral tumours: study protocol for a randomised controlled trial. BMJ Open. 2017 Nov 17;7(11):e018560. doi: 10.1136/bmjopen-2017-018560. PMID 29151054
- See also: Product resume on Phenylephrine — https://pro.medicin.dk/Medicin/Praeparater/3206
- See also: Product resume on Ephedrine — https://pro.medicin.dk/Medicin/Praeparater/3205